CLINICAL TRIAL: NCT02632006
Title: A Clinical Study of Adoptive Cellular Immunotherapy Using Pluripotent Killer T Cells Expressing Antibodies for Programmed Death 1 (PD-1) in Treating Patients With Advanced Hepatocellular Carcinoma
Brief Title: Immunotherapy Using Pluripotent Killer-Programmed Cell Death 1 (PIK-PD-1) Cells for the Treatment of Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2015-02-009
Record Dates: First submitted 2015-12-13; First posted 2015-12-16 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-09

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: PIK-PD-1 Cells; dendritic cell-precision multiple antigen T cells; advanced hepatocellular carcinoma

ARMS (2):
- PIK-PD-1 cells (Experimental): PIK-PD-1 cells treatment will be performed every 3 weeks with a total of three periods.
  Interventions: Biological: PIK-PD-1 cells
- DC-PMAT (Active Comparator): DC-PMAT cells treatment will be performed every 3 weeks with a total of three periods.
  Interventions: Biological: DC-PMAT

INTERVENTIONS:
Biological: PIK-PD-1 cells — DC cell suspension (1×10*7 DC+ physiological saline
  + 0.25% human serum albumin) 1ml for each infusion, subcutaneous injection for each infusion 3 cycles, each cycle received two infusions on day 19, 20; 40, 41; 61, 62. PIK-PD-1 cell suspension (1-6×10*9 PIK-PD-1 + physiological saline + 0.25% human serum albumin) 300ml for each infusion, IV (in the vein) for each infusion 3 cycles, each cycle received one infusions on day 21, 42, 63.
  Arms: PIK-PD-1 cells
Biological: DC-PMAT — DC cell suspension (1×10*7 DC+ physiological saline
  + 0.25% human serum albumin) 1ml for each infusion, subcutaneous injection for each infusion 3 cycles, each cycle received two infusions on day 19, 20; 40, 41; 61, 62. PMAT cell suspension (1-6×10*9 PMAT + physiological saline + 0.25% human serum albumin) 300ml for each infusion, IV (in the vein) for each infusion 3 cycles, each cycle received one infusions on day 21, 42, 63.
  Arms: DC-PMAT

SUMMARY:
Objectives:

The purpose of this study is to evaluate the safety and efficacy of PIK-PD-1 Cells in the treatment of advanced Hepatocellular Carcinoma.

Methods:

This study designs a novel therapy using PIK-PD-1 cells. 40 patients with advanced Hepatocellular Carcinoma will be enrolled. They are randomly divided into dendritic cell-precision multiple antigen T cells (DC-PMAT) group and PIK-PD-1 cells group. Both DC-PMAT treatment and PIK-PD-1 cells treatment will be performed every 3 weeks with a total of three periods. The mail clinical indicators are Progression-Free-Survival and Overall Survival.

DETAILED DESCRIPTION:
A total of 40 patients may be enrolled over a period of 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 20~70 years old, male or female; 2. Barcelona Clinic Liver Cancer(BCLC) C stage; no indication for operation, local treatment (Transcatheter Arterial Chemoembolization (TACE), percutaneous icro wave coagulation therapy (PMCT), percutaneous ethanol injection therapy (PEIT)) and radiation therapy; unable or unwilling to receive sorafenib therapy; 3.Child-Pugh score ≤ 9; 4.Eastern Cooperative Oncology Group (ECOG) score ≤ 2; 5.Life expectancy>3 months; 6. white blood cell (WBC) > 3 x 10*9/L, Neutrophils > 1 x 10*9/L, lymphocyte > 1 x 10*9/L, hemoglobin ≥8.5g/dl, Platelet ≥50×109/L, prothrombin time (PT) no more than 3 seconds, Cr and blood urea nitrogen (BUN) less than 3 times of the normal level; 7. Adequate venous access, blood cell production without other taboos; 8. Signed informed consent.

Exclusion Criteria:

* 1. Immunosuppressive therapy needed with autoimmune disease or organ transplantation history； 2. HIV/Syphilis infection; 3. Positive blood culture or imaging evidence infection; 4. Other drugs, gene therapy, biological, chemotherapy or radiation therapy were used within 1 months.

  5. The history of allergic reactions in cell therapy or cytokine. 6. PD-1 antibodies have been used before, or allergies due to PD-1 antibody drugs.

  7. History of interstitial lung disease. 8. History of esophagus varicosis rupture haemorrhage. 9. Other serious diseases:the heart,lung, kidney, digestive, nervous, mental disorders, immune regulatory diseases, metabolic diseases, infectious diseases, Etc.

  10. Pregnant, lactating women, or pregnancy planned at the following 2 years. 11. Without signed informed consent. 12. Other researchers considered ones unsuitable for inclusion.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 yeas

SECONDARY OUTCOMES:
Progress-free survival | 2 yeas
Quality of life | 2 yeas
  Quality of life core questionnaire will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Qijun Qian, PHD, Study Chair — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, China

REFERENCES:
- [Background] Cai XY, Gao Q, Qiu SJ, Ye SL, Wu ZQ, Fan J, Tang ZY. Dendritic cell infiltration and prognosis of human hepatocellular carcinoma. J Cancer Res Clin Oncol. 2006 May;132(5):293-301. doi: 10.1007/s00432-006-0075-y. Epub 2006 Jan 19. PMID 16421755
- [Background] Lee WC, Wang HC, Hung CF, Huang PF, Lia CR, Chen MF. Vaccination of advanced hepatocellular carcinoma patients with tumor lysate-pulsed dendritic cells: a clinical trial. J Immunother. 2005 Sep-Oct;28(5):496-504. doi: 10.1097/01.cji.0000171291.72039.e2. PMID 16113606
- [Background] Gonzalez-Carmona MA, Marten A, Hoffmann P, Schneider C, Sievers E, Schmidt-Wolf IG, Sauerbruch T, Caselmann WH. Patient-derived dendritic cells transduced with an a-fetoprotein-encoding adenovirus and co-cultured with autologous cytokine-induced lymphocytes induce a specific and strong immune response against hepatocellular carcinoma cells. Liver Int. 2006 Apr;26(3):369-79. doi: 10.1111/j.1478-3231.2005.01235.x. PMID 16584401
- [Background] Yannelli JR, Sturgill J, Foody T, Hirschowitz E. The large scale generation of dendritic cells for the immunization of patients with non-small cell lung cancer (NSCLC). Lung Cancer. 2005 Mar;47(3):337-50. doi: 10.1016/j.lungcan.2004.08.008. PMID 15713517
- [Background] Chang GC, Lan HC, Juang SH, Wu YC, Lee HC, Hung YM, Yang HY, Whang-Peng J, Liu KJ. A pilot clinical trial of vaccination with dendritic cells pulsed with autologous tumor cells derived from malignant pleural effusion in patients with late-stage lung carcinoma. Cancer. 2005 Feb 15;103(4):763-71. doi: 10.1002/cncr.20843. PMID 15637694
- [Background] Bellik L, Gerlini G, Parenti A, Ledda F, Pimpinelli N, Neri B, Pantalone D. Role of conventional treatments on circulating and monocyte-derived dendritic cells in colorectal cancer. Clin Immunol. 2006 Oct;121(1):74-80. doi: 10.1016/j.clim.2006.06.011. Epub 2006 Aug 17. PMID 16914380
- [Background] Babatz J, Rollig C, Lobel B, Folprecht G, Haack M, Gunther H, Kohne CH, Ehninger G, Schmitz M, Bornhauser M. Induction of cellular immune responses against carcinoembryonic antigen in patients with metastatic tumors after vaccination with altered peptide ligand-loaded dendritic cells. Cancer Immunol Immunother. 2006 Mar;55(3):268-76. doi: 10.1007/s00262-005-0021-x. Epub 2005 Jul 21. PMID 16034561
- [Background] Fay JW, Palucka AK, Paczesny S, Dhodapkar M, Johnston DA, Burkeholder S, Ueno H, Banchereau J. Long-term outcomes in patients with metastatic melanoma vaccinated with melanoma peptide-pulsed CD34(+) progenitor-derived dendritic cells. Cancer Immunol Immunother. 2006 Oct;55(10):1209-18. doi: 10.1007/s00262-005-0106-6. Epub 2005 Dec 6. PMID 16331519
- [Background] Davis ID, Chen Q, Morris L, Quirk J, Stanley M, Tavarnesi ML, Parente P, Cavicchiolo T, Hopkins W, Jackson H, Dimopoulos N, Tai TY, MacGregor D, Browning J, Svobodova S, Caron D, Maraskovsky E, Old LJ, Chen W, Cebon J. Blood dendritic cells generated with Flt3 ligand and CD40 ligand prime CD8+ T cells efficiently in cancer patients. J Immunother. 2006 Sep-Oct;29(5):499-511. doi: 10.1097/01.cji.0000211299.29632.8c. PMID 16971806
- [Background] Escobar A, Lopez M, Serrano A, Ramirez M, Perez C, Aguirre A, Gonzalez R, Alfaro J, Larrondo M, Fodor M, Ferrada C, Salazar-Onfray F. Dendritic cell immunizations alone or combined with low doses of interleukin-2 induce specific immune responses in melanoma patients. Clin Exp Immunol. 2005 Dec;142(3):555-68. doi: 10.1111/j.1365-2249.2005.02948.x. PMID 16297169
- [Background] Thomas-Kaskel AK, Zeiser R, Jochim R, Robbel C, Schultze-Seemann W, Waller CF, Veelken H. Vaccination of advanced prostate cancer patients with PSCA and PSA peptide-loaded dendritic cells induces DTH responses that correlate with superior overall survival. Int J Cancer. 2006 Nov 15;119(10):2428-34. doi: 10.1002/ijc.22097. PMID 16977630
- [Background] Fuessel S, Meye A, Schmitz M, Zastrow S, Linne C, Richter K, Lobel B, Hakenberg OW, Hoelig K, Rieber EP, Wirth MP. Vaccination of hormone-refractory prostate cancer patients with peptide cocktail-loaded dendritic cells: results of a phase I clinical trial. Prostate. 2006 Jun 1;66(8):811-21. doi: 10.1002/pros.20404. PMID 16482569
- [Background] Kyte JA, Gaudernack G. Immuno-gene therapy of cancer with tumour-mRNA transfected dendritic cells. Cancer Immunol Immunother. 2006 Nov;55(11):1432-42. doi: 10.1007/s00262-006-0161-7. Epub 2006 Apr 13. PMID 16612595
- [Background] Wang QJ, Hanada K, Perry-Lalley D, Bettinotti MP, Karpova T, Khong HT, Yang JC. Generating renal cancer-reactive T cells using dendritic cells (DCs) to present autologous tumor. J Immunother. 2005 Nov-Dec;28(6):551-9. doi: 10.1097/01.cji.0000175495.13476.1f. PMID 16224272
- [Background] Holtl L, Ramoner R, Zelle-Rieser C, Gander H, Putz T, Papesh C, Nussbaumer W, Falkensammer C, Bartsch G, Thurnher M. Allogeneic dendritic cell vaccination against metastatic renal cell carcinoma with or without cyclophosphamide. Cancer Immunol Immunother. 2005 Jul;54(7):663-70. doi: 10.1007/s00262-004-0629-2. Epub 2004 Dec 17. PMID 15918076
- [Background] Ferrari S, Malugani F, Rovati B, Porta C, Riccardi A, Danova M. Flow cytometric analysis of circulating dendritic cell subsets and intracellular cytokine production in advanced breast cancer patients. Oncol Rep. 2005 Jul;14(1):113-20. PMID 15944777
- [Background] Bohnenkamp HR, Coleman J, Burchell JM, Taylor-Papadimitriou J, Noll T. Breast carcinoma cell lysate-pulsed dendritic cells cross-prime MUC1-specific CD8+ T cells identified by peptide-MHC-class-I tetramers. Cell Immunol. 2004 Sep-Oct;231(1-2):112-25. doi: 10.1016/j.cellimm.2004.12.007. Epub 2005 Feb 8. PMID 15919376
- [Background] Chen W, Chan AS, Dawson AJ, Liang X, Blazar BR, Miller JS. FLT3 ligand administration after hematopoietic cell transplantation increases circulating dendritic cell precursors that can be activated by CpG oligodeoxynucleotides to enhance T-cell and natural killer cell function. Biol Blood Marrow Transplant. 2005 Jan;11(1):23-34. doi: 10.1016/j.bbmt.2004.08.004. PMID 15625541
- [Background] Triozzi PL, Khurram R, Aldrich WA, Walker MJ, Kim JA, Jaynes S. Intratumoral injection of dendritic cells derived in vitro in patients with metastatic cancer. Cancer. 2000 Dec 15;89(12):2646-54. doi: 10.1002/1097-0142(20001215)89:123.0.co;2-a. PMID 11135227
- [Background] Nestle FO. Dendritic cell vaccination for cancer therapy. Oncogene. 2000 Dec 27;19(56):6673-9. doi: 10.1038/sj.onc.1204095. PMID 11426654
- [Background] Mackensen A, Herbst B, Chen JL, Kohler G, Noppen C, Herr W, Spagnoli GC, Cerundolo V, Lindemann A. Phase I study in melanoma patients of a vaccine with peptide-pulsed dendritic cells generated in vitro from CD34(+) hematopoietic progenitor cells. Int J Cancer. 2000 May 1;86(3):385-92. doi: 10.1002/(sici)1097-0215(20000501)86:33.0.co;2-t. PMID 10760827
- [Background] Iinuma T, Homma S, Noda T, Kufe D, Ohno T, Toda G. Prevention of gastrointestinal tumors based on adenomatous polyposis coli gene mutation by dendritic cell vaccine. J Clin Invest. 2004 May;113(9):1307-17. doi: 10.1172/JCI17323. PMID 15124022
- [Background] Butterfield LH, Ribas A, Dissette VB, Amarnani SN, Vu HT, Oseguera D, Wang HJ, Elashoff RM, McBride WH, Mukherji B, Cochran AJ, Glaspy JA, Economou JS. Determinant spreading associated with clinical response in dendritic cell-based immunotherapy for malignant melanoma. Clin Cancer Res. 2003 Mar;9(3):998-1008. PMID 12631598
- [Background] Schuler-Thurner B, Schultz ES, Berger TG, Weinlich G, Ebner S, Woerl P, Bender A, Feuerstein B, Fritsch PO, Romani N, Schuler G. Rapid induction of tumor-specific type 1 T helper cells in metastatic melanoma patients by vaccination with mature, cryopreserved, peptide-loaded monocyte-derived dendritic cells. J Exp Med. 2002 May 20;195(10):1279-88. doi: 10.1084/jem.20012100. PMID 12021308
- [Background] O'Rourke MG, Johnson M, Lanagan C, See J, Yang J, Bell JR, Slater GJ, Kerr BM, Crowe B, Purdie DM, Elliott SL, Ellem KA, Schmidt CW. Durable complete clinical responses in a phase I/II trial using an autologous melanoma cell/dendritic cell vaccine. Cancer Immunol Immunother. 2003 Jun;52(6):387-95. doi: 10.1007/s00262-003-0375-x. Epub 2003 Apr 8. PMID 12682787